CLINICAL TRIAL: NCT02820285
Title: Characterization of Immune Semaphorin in Non Alcoholic Fatty Liver Disease and NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-PP-10
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2016-06

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Morbid obese patients (Other)
  Interventions: Other: Evaluation of the staging of fibrosis liver; Other: Determine the expression level of semaphorin; Other: Determination of the composition of immunity cells
- Control patients (Other)
  Interventions: Other: Evaluation of the staging of fibrosis liver; Other: Determine the expression level of semaphorin; Other: Determination of the composition of immunity cells
- Patients with overweight, steatosis and steatohepatitis (Other)
  Interventions: Other: Evaluation of the staging of fibrosis liver; Other: Determine the expression level of semaphorin; Other: Determination of the composition of immunity cells

INTERVENTIONS:
Other: Evaluation of the staging of fibrosis liver — The investigators will determine the severity of steatosis, inflammation and fibrosis by histological study of liver biopsies
Other: Determine the expression level of semaphorin — The investigators will determine the expression level (gene and protein) of immune semaphorin and their (s) receptor (s) in the liver and subcutaneous and visceral adipose tissue by RT-PCR,
Other: Determination of the composition of immunity cells — The investigators determine the composition of immunity cells by immunohistochemical and biochemical analyses (Western Blotting
  )

SUMMARY:
Recent epidemiological studies in France showed a high prevalence of obesity (14.5%) and its strong increase in the last 20 years. Among the many complications associated with obesity, liver complications (steatosis and steatohepatitis [NASH]) are among the most common. Semaphorins were described in the early 1990. More than 20 types of these proteins have been reported to date. These proteins were used for neural development. Since many functions have also been described. The semaphorins are involved in numerous physiological or physiopathological processes (cardiac morphogenesis, vascular growth, tumor progression), the regulation of immune cells and liver fibrosis. Preliminary studies have allowed to show that dendritic cells infiltrate adipose tissue and initiate the activation of T cells and inflammation. Immune semaphorin are new players in the regulation of inflammation and immune reactions.

The role of immune semaphorin in regulating inflammation in the two compartments (liver and adipose tissue) could be a crucial step that could lead to more severe liver damage. Its dysregulation could explain NASH injuries. The goal is to identify a new mode of regulation of cellular homeostasis in the fatty liver disease. These factors may serve as diagnostic markers or future therapeutic targets.

ELIGIBILITY:
Morbid obese patients

Inclusion Criteria:

* Male and female aged 18-65 years
* Patients with body mass index justifying a surgery for obesity (BMI ≥ 40 kg / m2 or BMI ≥ 35 kg / m2 with comorbidities)
* Consumption of alcohol <20 g / d
* Patients affiliated to a social security insurance
* Patients who signed the informed consent

Exclusion Criteria:

* Hemochromatosis
* Toxic hepatitis
* Deficiency of alpha-1-antitrypsin
* Wilson's disease
* Liver Autoimmune disease (primary biliary cirrhosis, autoimmune hepatitis)
* Hepatitis B, C
* Drug-induced hepatitis
* Presence of HIV status
* Corticosteroids, amiodarone, valproic acid, tamoxifen, anti-inflammatory drugs, lipid lowering agents, testosterone agonists or beta-adrenergic antagonists, orlistat.
* Pregnant or breastfeeding women
* Incarcerated patients or patient under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the staging of liver fibrosis | Day 0
  The investigators determine the stage of liver fibrosis by histological study of biopsies
Determination of the expression of level of semaphorin | Day 0
  The investigators determine by technic of Reverse Transcription Polymerase Chain Reaction (RT-PCR) the expression of level of semaphorin
Determination of the composition of immunity cells | Day 0
  The investigators determine the composition of immunity cells by Immunohistochemical and biochemical analyses (Western Blotting)

CONTACTS AND LOCATIONS:
Overall Officials: Albert TRAN, MDPhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Service d'Hépato-Gastroentérologie - Hôpital de l'Archet, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sans A, Bailly L, Anty R, Sielezenef I, Gugenheim J, Tran A, Gual P, Iannelli A. Baseline Anthropometric and Metabolic Parameters Correlate with Weight Loss in Women 1-Year After Laparoscopic Roux-En-Y Gastric Bypass. Obes Surg. 2017 Nov;27(11):2940-2949. doi: 10.1007/s11695-017-2720-8. PMID 28550439